CLINICAL TRIAL: NCT02617849
Title: A Phase II Study of Pembrolizumab With Carboplatin/Paclitaxel in Patients With Metastatic Melanoma
Brief Title: Pembrolizumab With Carboplatin/Paclitaxel in Patients With Metastatic Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wilson Miller (Other)
Responsible Party: Sponsor-Investigator, Wilson Miller, Medical Oncologist, Jewish General Hospital
Organization: Jewish General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-3475-269
Record Dates: First submitted 2015-11-03; First posted 2015-12-01 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Metastatic Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pembrolizumab, Carboplatin, Paclitaxel (Experimental): Carboplatin will be administered at AUC = 6, IV over 60 minutes every 3 weeks for up to 4 doses. Paclitaxel will be administered at 175mg/m2, IV over 3 hours every 3 weeks for up to 4 doses. Pembrolizumab will be administered at 200 mg, IV over 30 minutes every 3 weeks.
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg IV every 3 weeks
  Other Names: MK3475
Drug: Carboplatin — AUC=6, every 3 weeks x 4
Drug: Paclitaxel — 175 mg/m2, every 3 weeks x 4

SUMMARY:
This is a multi-center, open-label, Phase II clinical trial evaluating pembrolizumab in combination with carboplatin/paclitaxel as a treatment in unresectable locally advanced or metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

The subject must:

1. Be willing and able to provide written informed consent for the trial.
2. Be ≥ 18 years of age on day of signing informed consent.
3. Have histologically confirmed diagnosis of unresectable Stage III or metastatic melanoma.

   * Patients may not have a diagnosis of uveal melanoma.
4. Have measurable disease based on RECIST 1.1.
5. Have a tumor sample (FFPE archival or newly obtained biopsy) of a metastatic site that is available for biomarker analysis.
6. Have an ECOG of 0 or 1.
7. Demonstrate adequate organ function as below:

   * Absolute neutrophil count (ANC) ≥1.5 x 109/L
   * Platelets ≥100 x 109/L
   * Hemoglobin ≥90 g/L (may be transfused)
   * Serum creatinine OR CrCl ≤ 1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
   * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
   * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
   * Albumin >2.5 mg/dL
   * International Normalized Ratio (INR) or Prothrombin Time (PT)
   * Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
10. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
11. No known active or chronic infection with HIV, Hepatitis B, or Hepatitis C.

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

1. Has had prior treatment for advanced unresectable or metastatic melanoma. Prior treatment with BRAF and MEK inhibitors is permitted in this setting. A washout of at least 5-half-lives (median terminal half-life) prior to the first dose of trial treatment must have elapsed.
2. Has received prior therapy with an anti-CTLA4, anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
3. Has evidence of symptomatic CNS lesions as determined by the investigator. Patients with asymptomatic lesions or previously irradiated or surgically resected are eligible.
4. Has a known additional malignancy that is progressing or requires active treatment.
5. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (>10 mg daily prednisone equivalents) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Inhaled or topical steroids, and adrenal replacement doses ≤ 10 mg prednisone equivalents are permitted.
6. Has ≥ Grade 2 peripheral neuropathy.
7. Patients with an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents. Patients with vitiligo or resolved childhood asthma/atopy is an exception to this rule. Patients that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Patients with hypothyroidism stable on hormone replacement will not be excluded from the study.
8. Has an active infection requiring systemic therapy.
9. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
10. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
11. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
12. Has a known history of active TB (Bacillus Tuberculosis)
13. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate as assessed by RECIST 1.1 and immune-related Response Criteria | 56 months

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 56 months
Overall Survival | 56 months
Progression Free Survival | 56 months
Melanoma-associated serological markers by multiplexed array will be generated | 56 months

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Miller, MD, PhD, Principal Investigator — Jewish General Hospital; Rahima Jamal, MD, PhD, Principal Investigator — CHUM, Hopital Notre-Dame
Locations (2):
- Canada (2):
  - Jewish General Hospital, Montreal, Quebec
  - Hopital Notre-Dame, Montreal, Quebec